CLINICAL TRIAL: NCT02919397
Title: Effectiveness of Integrating Motivational Instant Messaging Into an E-diabetes Prevention Programme in People at High Risk of Type 2 Diabetes: a Prospective, Parallel-group, Randomised Controlled Trial (Diabetes Stopwatch)
Brief Title: Motivational Instant Messaging and E-diabetes Prevention Programme for High Risk of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 197384
Record Dates: First submitted 2016-09-20; First posted 2016-09-29 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-03

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Wearable Electronic Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): If participants are allocated to the intervention group, participants will receive the wearable technology and access to the smartphone application. Motivational messages based on diabetes prevention programme content, and biofeedback messages based on physical activity data provided via the wearable technology, will be received by participants via the application. The diabetes prevention programme educational material will be available via the application.
  Interventions: Device: Wearable technology; Behavioral: Diabetes Prevention Programme educational material; Behavioral: Motivational messaging
- Control (Active Comparator): If participants are allocated to the control group, participants will receive the wearable technology and will be able to access their activity data via the smartphone application. Participants will also have have access to the diabetes prevention programme educational material via the application. Participants will not receive motivational messages related to the education content or activity data.
  Interventions: Device: Wearable technology; Behavioral: Diabetes Prevention Programme educational material

INTERVENTIONS:
Device: Wearable technology — Buddi wearable technology will record activity levels, participants will access activity data through smartphone application
Behavioral: Diabetes Prevention Programme educational material — Educational material accessed through smartphone application
Behavioral: Motivational messaging — Messages sent via smartphone application
  Arms: Intervention

SUMMARY:
The overall aim of this feasibility trial is to assess the effectiveness of a wearable technology and an e-diabetes prevention programme delivered via a smartphone application, including motivational messaging, in reducing weight and increasing physical activity in people at risk of developing type 2 diabetes.

DETAILED DESCRIPTION:
The study will examine whether a wearable technology, combined with biofeedback, motivational messaging and an e-diabetes prevention programme, is effective in reducing weight and increasing physical activity after 12 months.

The intervention will consist of a wearable technology and a smartphone application made available for a 12 month period. 22 online multimedia sessions targeting diet, physical activity and mental resilience delivered via the smartphone application. Motivational messaging based on the diabetes prevention module content and biofeedback will be sent to participants via the application.

The control group will receive the wearable technology and will have access to a smartphone application detailing their activity. Participants will be directed to the same educational material as is made available via the multimedia sessions, but will not receive motivational messages.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c between 42 and 47 mmol/mol
* BMI≥25 kg/m²
* Fluent in conversational English
* Permanent resident in Lambeth, Southwark or Lewisham
* Ownership of a smartphone (iPhone or Android only) for communication defined as logging on at least once/day to the internet
* Ambulatory.

Exclusion Criteria:

* Known diabetes
* Pregnancy or planning pregnancy during the duration of the study
* Severe mental illness (severe depression, psychosis, bipolar affective disorder, dementia, learning difficulties, substance problem use or dependence)
* Severe physical disability e.g. that would prevent any increased uptake of physical exercise
* Advanced active disease such as cancer or heart failure
* Any other condition which requires glucose altering drugs
* Morbid obesity (BMI ≥50 kg/m²)
* Current participation in a weight loss programme.

When in doubt the investigators will seek the GP opinion and approval.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Physical activity (average steps per day) | 7 days
  Average steps taken per day from 7 days wear measured using the Buddi wearable technology, which will be worn 24 hours per day for 7 days
Weight (kg) | At 12 month follow-up appointment
  Measured in light clothing, without shoes, on the a Class 3 Tanita SC240 weighing digital scale to 0.01 kg for weight

SECONDARY OUTCOMES:
HbA1c (mmol/mol) | At 12 month follow-up appointment
Height (cm) | At 12 month follow-up appointment
BMI (kg/m^2) | At 12 month follow-up appointment
Waist circumference (cm) | At 12 month follow-up appointment
Hip circumference (cm) | At 12 month follow-up appointment
Total cholesterol (mmol/L) | At 12 month follow-up appointment
High density lipoprotein cholesterol (mmol/L) | At 12 month follow-up appointment
Low density lipoprotein cholesterol (mmol/L) | At 12 month follow-up appointment
Systolic blood pressure (mmHg) | At 12 month follow-up appointment
Diastolic blood pressure (mmHg) | At 12 month follow-up appointment
Sleep duration (average hours per night) | 7 days
  The Buddi wearable technology will be worn for 24 hours per day. Therefore, during sleeping hours participant activity will be measured and duration of sleep can be calculated. Participants will wear the Buddi device for 7 days, and the average number of hours sleep per night will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Khalida Ismail, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Staite E, Bayley A, Al-Ozairi E, Stewart K, Hopkins D, Rundle J, Basudev N, Mohamedali Z, Ismail K. A Wearable Technology Delivering a Web-Based Diabetes Prevention Program to People at High Risk of Type 2 Diabetes: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 15;8(7):e15448. doi: 10.2196/15448. PMID 32459651